Cover Page: Statistical Analysis Plan We The Village Counselor Training Study

NCT05875142

Document Date: 09.26.23

## **Statistical Analysis Plan**

Our statistical analysis focuses on a primary endpoint as well as a number of secondary endpoints of interest. The data derive from questionnaires collected from participants in the study. The final enrollment involved three groups: T – Digital Tutorial Overview, TM – Digital Tutorial Plus Training Materials, and TMC – Digital Tutorial Plus Training Materials Plus Feedback and Coaching, with 15, 16, and 16 subjects enrolled, respectively.

- 1. T Digital Tutorial Overview: Participants assigned to T were given access to a digital tutorial consisting of a curriculum dashboard for review of 10 modules, including videos, PDFs, text and quizzes, which are to be self-administered over two weeks. Modules remain available during the 10-week post tutorial period. Participants receive weekly contact encouraging engagement in all of the materials available to them.
- 2. TM Digital Tutorial Plus Training Materials: Participants receive the digital tutorial (T) as described above plus access to 10 modules of digital training materials released weekly over the 10-week post tutorial period for self-study. Participants receive weekly contact encouraging engagement in all of the materials available to them.
- 3. TMC Digital Tutorial Plus Training Materials Plus Feedback and Coaching:

  Participants receive the digital tutorial (T) plus the digital Training materials as described in the two arms above plus they submit audio recordings of sessions with clients and receive feedback on their application of CRAFT and coaching on how to improve. Participants receive weekly contact encouraging engagement in all of the materials available to them.

Our comparisons are all treatment/control comparisons of T with TM, and T with TMC.

## 1. Primary Hypothesis

1.1. At 12 weeks (after study start), participants assigned to the TMC condition will demonstrate the highest CRAFT procedure fidelity (measured in audiotaped sessions with a standardized patient) followed by TM and then T. *Rationale*: Direct observation measuring content of CRAFT delivered in treatment sessions is our primary outcome as this provides the best assessment of counselor adherence and skill and is consistent with previous studies.<sup>7,10,41</sup> Our hypothesis that TMC will produce greater use of CRAFT than T (or TM) is based on the results from previous trials comparing a workshop only to workshops plus feedback and coaching.<sup>7,10,41</sup>

## 2. Secondary Hypotheses

- 2.1. Participants assigned to the TMC condition will demonstrate the highest CRAFT knowledge followed by TM and then T, in their 12-week knowledge test.

  <u>Rationale</u>: Results from previous controlled trials have shown no differences in counselor knowledge pre- to post-workshop, but increases have been seen when fact sheets and supervision are added after the workshop.<sup>39,57-58</sup>
- 2.2. Participants in all conditions will perceive increased implementation potential over time (pre-tutorial, post-tutorial, 12 week follow up), but at 12 weeks implementation potential will be lower for TMC compared to TM and T.
  <u>Rationale</u>: In a CBT (Cognitive Behavioral Therapy) web-based training study implementation potential of three training programs increased over time, but a condition involving expert supervision was seen as more difficult to implement.<sup>39</sup>

2.3. Participants assigned to the TMC condition will report that more IPs have entered treatment compared to TM and T at 12-weeks (after study start) follow-up surveys. *Rationale*: This hypothesis is based on the results from previous trials examining counselor fidelity <sup>7,10,41</sup> and studies showing that CBT fidelity enhances treatment outcome. <sup>59-60</sup> We consider this hypothesis exploratory because the 6 month timeline will not be sufficient to adequately test for differences in treatment entry, as there would not be much time after all counselors completed training for them to complete CRAFT with CSOs.

## Data Analysis

Primary and secondary hypotheses were investigated by computing the improvement from baseline to 12-week timepoints. One-sided independent samples T-tests were used for pairwise comparisons of the three conditions. One-sided tests are appropriate for our hypothesized conditions: the alternative hypotheses for which we seek evidence is TMC is better than T, TM is better than T, and TMC is better than TM.